CLINICAL TRIAL: NCT00413283
Title: Phase 2, Randomized, Double Blind, Placebo-Controlled Dose and Schedule Finding Trial to Evaluate the Safety and Efficacy of AMG 531 For Treatment of Chemotherapy-Induced Thrombocytopenia in Subjects With Advanced Non-Small Cell Lung Cancer Already Receiving Gemcitabine and Platinum.
Brief Title: Dose/ Schedule Finding Trial of Romiplostim for Chemotherapy-Induced Thrombocytopenia (CIT) in Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20050154
Record Dates: First submitted 2006-12-15; First posted 2006-12-19 (Estimated); Results first posted 2010-10-21 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-09

CONDITIONS: Lung Cancer; Chemotherapy-Induced Thrombocytopenia; Non-Small Cell Lung Cancer; Cancer; Lung Neoplasms; Oncology; Solid Tumors; Thrombocytopenia
Keywords: Advanced Non-Small Cell Lung Cancer; Chemotherapy Induced Thrombocytopenia; CIT; NSCLC; Stage IIIB NSCLC; Stage IV NSCLC; Gemcitabine; Carboplatin; Cisplatin
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms; Thrombocytopenia | interventions — romiplostim; Gemcitabine; Carboplatin; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): Participants received a placebo subcutaneous injection on Day 2 of each chemotherapy cycle. Chemotherapy consisted of 21-day cycles of gemcitabine/carboplatin (gemcitabine and carboplatin on Day 1 and gemcitabine again on Day 8) or 21-day cycles of gemcitabine/cisplatin (gemcitabine and cisplatin on Day 1 and gemcitabine again on Day 8), up to a maximum of 5 cycles administered according to standard institutional practice.
  Interventions: Drug: Placebo; Drug: Gemcitabine; Drug: Carboplatin; Drug: Cisplatin
- Romiplostim 250 μg (Experimental): Participants received romiplostim 250 μg administered subcutaneously on Day 2 of each chemotherapy cycle. Chemotherapy consisted of 21-day cycles of gemcitabine/carboplatin (gemcitabine and carboplatin on Day 1 and gemcitabine again on Day 8) or 21-day cycles of gemcitabine/cisplatin (gemcitabine and cisplatin on Day 1 and gemcitabine again on Day 8), up to a maximum of 5 cycles administered according to standard institutional practice.
  Interventions: Biological: Romiplostim; Drug: Gemcitabine; Drug: Carboplatin; Drug: Cisplatin
- Romiplostim 500 μg (Experimental): Participants received romiplostim 500 μg administered subcutaneously on Day 2 of each chemotherapy cycle. Chemotherapy consisted of 21-day cycles of gemcitabine/carboplatin (gemcitabine and carboplatin on Day 1 and gemcitabine again on Day 8) or 21-day cycles of gemcitabine/cisplatin (gemcitabine and cisplatin on Day 1 and gemcitabine again on Day 8), up to a maximum of 5 cycles administered according to standard institutional practice.
  Interventions: Biological: Romiplostim; Drug: Gemcitabine; Drug: Carboplatin; Drug: Cisplatin
- Romiplostim 750 μg (Experimental): Participants received romiplostim 750 μg administered subcutaneously on Day 2 of each chemotherapy cycle. Chemotherapy consisted of 21-day cycles of gemcitabine/carboplatin (gemcitabine and carboplatin on Day 1 and gemcitabine again on Day 8) or 21-day cycles of gemcitabine/cisplatin (gemcitabine and cisplatin on Day 1 and gemcitabine again on Day 8), up to a maximum of 5 cycles administered according to standard institutional practice.
  Interventions: Biological: Romiplostim; Drug: Gemcitabine; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Biological: Romiplostim — Romiplostim is a thrombopoiesis recombinant protein that targets the thrombopoietin (TPO) receptor which results in increased platelet production.
  Other Names: AMG 531; Nplate®
  Arms: Romiplostim 250 μg; Romiplostim 500 μg; Romiplostim 750 μg
Drug: Placebo — Placebo subcutaneous injection.
  Arms: Placebo
Drug: Gemcitabine — Intravenous infusion
Drug: Carboplatin — Intravenous infusion
Drug: Cisplatin — Intravenous infusion

SUMMARY:
The purpose of this study is to identify an effective, well tolerated dose and schedule of romiplostim that is appropriate for the treatment of chemotherapy induced thrombocytopenia (CIT) in patients with non-small cell lung cancer receiving gemcitabine and platinum.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic stage IIIB or stage IV NSCLC receiving 21-day cycles of gemcitabine/carboplatin or gemcitabine/cisplatin
* Life expectancy ≥ 12 weeks at the time of screening
* Thrombocytopenia as evidenced by a platelet count ≤ 50 x 10^9/L during the qualifying cycle of chemotherapy, OR platelet count < 100 x 10^9/L on Day 22 of the qualifying cycle (for eligibility inclusion: ability to receive the same dose of chemotherapy on study), this criteria ensures that the patient must be dose delayed for platelet recovery
* Ability to receive the same dose and schedule of chemotherapy during the first on-study treatment cycle as was given in the qualifying cycle (except Day 8 gemcitabine)
* Absolute neutrophil count (ANC) ≥ 1,000/µL, hemoglobin ≥ 9.5 g/dL, and platelet count ≥ 100 x 10 ^9/L on Day 1 of the first on study chemotherapy treatment cycle
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at the time of screening
* Adequate Liver function; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3.0 x upper limit of normal (ULN) (except for patients with a confirmed diagnosis of Gilbert's Syndrome)
* Adequate renal function; serum creatinine < 1.5 x ULN

Exclusion Criteria:

* Receipt of > 1 prior systemic chemotherapy regimen
* Sepsis, disseminated coagulation or any other condition (i.e. immune [idiopathic] thrombocytopenic purpura [ITP], thrombotic thrombocytopenic purpura [TTP], hemolytic uremic syndrome [HUS]) that may exacerbate thrombocytopenia
* History of unstable angina, congestive heart failure, uncontrolled hypertension (diastolic > 100 mmHg), uncontrolled cardiac arrhythmia, or recent (within 1 year of screening ) myocardial infarction
* History of arterial thrombosis (e.g., stroke or transient ischemic attack) within 1 year of screening
* History of pulmonary embolism or other venous thrombosis within 1 year of screening (except for catheter-related clots)
* Use of any nitrosourea or mitomycin-C within 6 weeks of screening
* Have received any thrombopoietic growth factor or related substance
* Have received granulocyte macrophage colony stimulating factor (GM-CSF) within the last 4 weeks prior to screening
* Have received any experimental therapy within 4 weeks prior to screening
* Have ever received a bone marrow or peripheral blood stem cell infusion (within 1 year of screening)
* Known hypersensitivity to any recombinant E. coli-derived product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (55):
- United States (25):
  - Research Site, Glendale, Arizona
  - Research Site, Anaheim, California
  - Research Site, Los Angeles, California
  - Research Site, Rancho Mirage, California
  - Research Site, Boynton Beach, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Athens, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Peoria, Illinois
  - Research Site, Sioux City, Iowa
  - Research Site, Paducah, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Sterling Heights, Michigan
  - Research Site, Billings, Montana
  - Research Site, Flemington, New Jersey
  - Research Site, Johnson City, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Drexel Hill, Pennsylvania
  - Research Site, Dunmore, Pennsylvania
  - Research Site, Radnor, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Germantown, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
- Austria (6):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Klagenfurt
  - Research Site, Linz
  - Research Site, Rankweil
  - Research Site, Vienna
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Sainte-Foy, Quebec
- Germany (4):
  - Research Site, Bad Berka
  - Research Site, Dresden
  - Research Site, Halle
  - Research Site, Hemer
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Edelény
  - Research Site, Gyula
  - Research Site, Mátraháza
  - Research Site, Pécs
  - Research Site, Székesfehérvár
  - Research Site, Törökbálint
  - Research Site, Zalaegerszeg - Pozva
- Ireland (2):
  - Research Site, Cork
  - Research Site, Dublin
- Italy (4):
  - Research Site, Novara
  - Research Site, Orbassano
  - Research Site, Palermo
  - Research Site, Torino
- Portugal (4):
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 28 December 2006 through 11 August 2008.
Groups:
- Romiplostim 250 µg: Participants received romiplostim 250 μg administered subcutaneously on Day 2 of each chemotherapy cycle. Chemotherapy consisted of 21-day cycles of gemcitabine/carboplatin (gemcitabine and carboplatin on Day 1 and gemcitabine again on Day 8) or 21-day cycles of gemcitabine/cisplatin (gemcitabine and cisplatin on Day 1 and gemcitabine again on Day 8), up to a maximum of 5 cycles administered according to standard institutional practice.
- Romiplostim 500 µg: Participants received romiplostim 500 μg administered subcutaneously on Day 2 of each chemotherapy cycle. Chemotherapy consisted of 21-day cycles of gemcitabine/carboplatin (gemcitabine and carboplatin on Day 1 and gemcitabine again on Day 8) or 21-day cycles of gemcitabine/cisplatin (gemcitabine and cisplatin on Day 1 and gemcitabine again on Day 8), up to a maximum of 5 cycles administered according to standard institutional practice.
- Romiplostim 750 µg: Participants received romiplostim 750 μg administered subcutaneously on Day 2 of each chemotherapy cycle. Chemotherapy consisted of 21-day cycles of gemcitabine/carboplatin (gemcitabine and carboplatin on Day 1 and gemcitabine again on Day 8) or 21-day cycles of gemcitabine/cisplatin (gemcitabine and cisplatin on Day 1 and gemcitabine again on Day 8), up to a maximum of 5 cycles administered according to standard institutional practice.
Period: Overall Study
Arm/Group | Placebo | Romiplostim 250 µg | Romiplostim 500 µg | Romiplostim 750 µg
Started | 12 | 16 | 18 | 17
Received Study Drug | 12 | 16 | 18 | 16
Completed | 11 | 13 | 16 | 13
Not Completed | 1 | 3 | 2 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Ineligibility determined | 0 | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 1 | 0 | 0
Not completed — Requirement for alternative therapy | 0 | 2 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romiplostim 250 µg | Romiplostim 500 µg | Romiplostim 750 µg | Total
Number analyzed (Participants) | 12 | 16 | 18 | 17 | 63
Age Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (6.6) | 63.8 (10.8) | 62.5 (7.7) | 65.4 (8.2) | 63.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 6 | 2 | 18
  Male | 6 | 12 | 12 | 15 | 45
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 12 | 15 | 18 | 17 | 62
  Black or African American | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: This summary includes all treatment-emergent adverse events recorded from the start of investigational product on this study, or any worsening of adverse events initially experienced before initiation of this study.
Time Frame: 4 months
Population: Safety Analysis Set, composed of all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo | Romiplostim 250 µg | Romiplostim 500 µg | Romiplostim 750 µg
Number analyzed (Participants) | 12 | 16 | 18 | 16
Participants | 12 | 16 | 18 | 14

2. Secondary Outcome: Duration of Grade 3 or 4 Thrombocytopenia
Description: The duration of grade 3 or 4 thrombocytopenia (defined as platelet count <50 x 10^9/L) experienced during the first on study chemotherapy cycle by treatment group.
Time Frame: 3 weeks
Population: Efficacy Analysis Set, composed of all randomized participants except those who were replaced (participants who discontinued prior to the completion of at least 1 romiplostim treatment cycle for non-platelet-related reasons).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Romiplostim 250 µg | Romiplostim 500 µg | Romiplostim 750 µg
Number analyzed (Participants) | 12 | 15 | 18 | 16
days | 2.1 (3.3) | 3.6 (4.3) | 2.6 (3.9) | 2.1 (2.7)
Statistical Analysis 1: Comparison: Placebo vs Romiplostim 750 µg; Test type: Superiority or Other; p = 0.972, Satterthwaite t-test
Statistical Analysis 2: Comparison: Placebo vs Romiplostim 500 µg; Test type: Superiority or Other; p = 0.725, Satterthwaite t-test
Statistical Analysis 3: Comparison: Placebo vs Romiplostim 250 µg; Test type: Superiority or Other; p = 0.312, Satterthwaite t-test

3. Secondary Outcome: Number of Participants Experiencing Grade 3 or 4 Thrombocytopenia During the First Treatment Cycle.
Description: The number of participants in each treatment group with grade 3 or 4 thrombocytopenia during the first on study treatment cycle. Per the Common Terminology Criteria for Adverse Events (CTCAE) v3.0, participants with a platelet count < 50 x 10^9/L, but ≥ 25 x 10^9/L are considered to have Grade 3 thrombocytopenia and participants with a platelet count < 25 x 10^9/L are considered to have Grade 4 thrombocytopenia. Additionally, participants with a platelet transfusion during the first on-study treatment cycle were classified as having Grade 3/4 thrombocytopenia.
Time Frame: 3 weeks
Population: Efficacy Analysis Set, composed of all randomized participants except those who were replaced.
Measure: Number; unit: Participants
Arm/Group | Placebo | Romiplostim 250 µg | Romiplostim 500 µg | Romiplostim 750 µg
Number analyzed (Participants) | 12 | 15 | 18 | 16
Participants | 5 | 7 | 7 | 7
Statistical Analysis 1: Comparison: Placebo vs Romiplostim 750 µg; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Romiplostim 500 µg; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs Romiplostim 250 µg; Test type: Superiority or Other; p = 1.000, Fisher Exact

4. Secondary Outcome: Number of Participants With Platelet Transfusions
Description: Number of participants who were administered platelet transfusions during first on study treatment cycle.
Time Frame: 3 weeks
Population: Efficacy Analysis Set, composed of all randomized participants except those who were replaced.
Measure: Number; unit: Participants
Arm/Group | Placebo | Romiplostim 250 µg | Romiplostim 500 µg | Romiplostim 750 µg
Number analyzed (Participants) | 12 | 15 | 18 | 16
Participants | 1 | 4 | 1 | 1
Statistical Analysis 1: Comparison: Placebo vs Romiplostim 750 µg; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Romiplostim 500 µg; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs Romiplostim 250 µg; Test type: Superiority or Other; p = 0.342, Fisher Exact

5. Secondary Outcome: Platelet Count on Day 22
Description: Platelet count on Day 22 of the first on study chemotherapy treatment cycle (planned Day 1 of next cycle) by treatment group
Time Frame: Day 22
Population: Efficacy Analysis Set, composed of all randomized participants except those who were replaced
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Placebo | Romiplostim 250 µg | Romiplostim 500 µg | Romiplostim 750 µg
Number analyzed (Participants) | 12 | 15 | 18 | 16
10^9/L | 281.2 (116.0) | 222.6 (112.0) | 412.8 (295.2) | 336.0 (254.9)
Statistical Analysis 1: Comparison: Placebo vs Romiplostim 750 µg; Test type: Superiority or Other; p = 0.454, Satterthwaite t-test
Statistical Analysis 2: Comparison: Placebo vs Romiplostim 500 µg; Test type: Superiority or Other; p = 0.101, Satterthwaite t-test
Statistical Analysis 3: Comparison: Placebo vs Romiplostim 250 µg; Test type: Superiority or Other; p = 0.199, Satterthwaite t-test

6. Secondary Outcome: Gemcitabine Dose Reduction on Day 8 of the First Chemotherapy Cycle
Description: Number of participants who required a gemcitabine dose reduction on Day 8 of the first on study chemotherapy cycle.
Time Frame: 8 days
Population: Efficacy Analysis Set, composed of all randomized participants except those who were replaced.
Measure: Number; unit: Participants
Arm/Group | Placebo | Romiplostim 250 µg | Romiplostim 500 µg | Romiplostim 750 µg
Number analyzed (Participants) | 12 | 15 | 18 | 16
Participants | 2 | 4 | 4 | 5
Statistical Analysis 1: Comparison: Placebo vs Romiplostim 750 µg; Test type: Superiority or Other; p = 0.662, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Romiplostim 500 µg; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs Romiplostim 250 µg; Test type: Superiority or Other; p = 0.662, Fisher Exact

ADVERSE EVENTS:
Time Frame: From signing of the informed consent through 30 days after the last dose of investigational product or end of study, whichever is longer (up to 4 months).
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo | Romiplostim 250 µg | Romiplostim 500 µg | Romiplostim 750 µg
Serious Adverse Events (participants affected / at risk) | 1/12 | 7/16 | 5/18 | 5/16
Other Adverse Events (participants affected / at risk) | 12/12 | 16/16 | 17/18 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Romiplostim 250 µg (N=16) | Romiplostim 500 µg (N=18) | Romiplostim 750 µg (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Romiplostim 250 µg (N=16) | Romiplostim 500 µg (N=18) | Romiplostim 750 µg (N=16)
Anaemia (Blood and lymphatic system disorders) | 6 | 7 | 7 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 4 | 4 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 5
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 8 | 8 | 8
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 5 | 2
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 4 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 1 | 1
Catheter site swelling (General disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 1
Face oedema (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 5 | 4 | 1
Infusion site extravasation (General disorders) | 0 | 1 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 2
Pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 5 | 2 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Fungal oesophagitis (Infections and infestations) | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 2 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 3
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 4 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 1 | 0
Phlebitis superficial (Vascular disorders) | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.